CLINICAL TRIAL: NCT03012048
Title: Effectiveness of Low-cost Point-of-use Water Treatment Technologies to Prevent Stunting Among Children in Limpopo, South Africa
Brief Title: Effectiveness of Point-of-use Water Treatment Technologies to Prevent Stunting Among Children in South Africa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: University of Venda (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB-HSR 18662
Record Dates: First submitted 2017-01-03; First posted 2017-01-06 (Estimated); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Diarrhoea;Infectious;Presumed; Diarrhea, Infantile; Diarrhea Tropical; Environmental Exposure; Enteropathy; Malnutrition, Child
Keywords: water treatment
MeSH Terms: conditions — Diarrhea, Infantile; Sprue, Tropical; Intestinal Diseases; Child Nutrition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- MadiDrop (ceramic tablet) (Experimental): Households receive a MadiDrop (silver-impregnated ceramic tablet) in a safe-storage water container to use for all drinking water needs in the household. MadiDrops are replaced every 6 months over the 2-year intervention study period.
  In July 2017, all households in the MadiDrop arm were crossed over to the ceramic water filter arm due to inconsistent silver release from the ceramic tablets.
  Interventions: Device: Silver-impregnated ceramic tablet
- Silver-impregnated ceramic water filter (Active Comparator): Households receive a silver-impregnated ceramic filter in a safe-storage water container to use for all drinking water needs in the household. Filters are replaced at the end of the 2-year intervention study period.
  In December 2017, all silver-impregnated ceramic water filters were replaced with the same ceramic filters without silver due to continued inconsistencies with silver release.
  Interventions: Device: Silver-impregnated ceramic water filter
- Safe-storage water container (Active Comparator): Households receive a safe-storage water container alone to use for all drinking water needs in the household.
  Interventions: Device: Safe-storage water container
- No intervention (No Intervention): Households are encouraged to continue their usual water treatment practices.

INTERVENTIONS:
Device: Silver-impregnated ceramic tablet — A silver-impregnated ceramic disk used for drinking water treatment that was developed by engineers at the University of Virginia. When the ceramic disk is placed in a household water storage container, silver diffuses through the porous ceramic into the water at a release rate that is effective for continual disinfection of waterborne pathogens while remaining below the silver drinking water standard. The disk is effective for daily treatment of 10 to 15 liters for at least six months.
  This intervention was removed from the study in July 2017 (approximately at 1 year of follow-up).
  Other Names: MadiDrop (trade name)
  Arms: MadiDrop (ceramic tablet)
Device: Silver-impregnated ceramic water filter — Silver-impregnated ceramic water filter are well-developed, tested, and widely-used devices. In addition to mechanically removing pathogens, the filter is treated with silver to reduce live pathogens that pass through the filter and to provide residual disinfectant to reduce risk of recontamination after treatment.
  This intervention was replaced with ceramic filters without silver in Dec 2017 (approximately at 1.5 years of follow-up).
  Arms: Silver-impregnated ceramic water filter
Device: Safe-storage water container — The safe-storage water containers used in this study are plastic buckets with a spigot, purchased locally.
  Arms: Safe-storage water container

SUMMARY:
This project is a community-based randomized controlled trial designed to test the effectiveness of two point-of-use water treatment technologies to improve clean drinking water access, reduce enteropathogen burden, and improve child growth among children in Limpopo, South Africa.

DETAILED DESCRIPTION:
Lack of access to safe water in low-resource settings likely contributes to stunted growth early in life, which affects more than a quarter of children under 5 years worldwide. Point-of-use water treatment technologies have the potential to provide effective and low-cost solutions to improving quality of drinking water in these settings. One such technology, a silver-impregnated ceramic disk, continually disinfects water in household water storage containers by diffusing silver into the water for daily treatment of 10 to 15 liters for at least six months. Silver-impregnated ceramic water filters are another commercially available technology that additionally remove pathogens mechanically. While both technologies have proven to be highly effective in treating water, it is unknown whether the use of these technologies will translate to improvements in child health outcomes. This community-based intervention trial will estimate the effect of the silver-impregnated ceramic disk and a silver-impregnated ceramic water filter on linear growth of children in Limpopo, South Africa.

Households in the Dzimauli community will be randomized to receive the ceramic disk, a water filter, the safe-storage water container alone, or no intervention. Children will be followed every three months for 2 years to assess height, weight, and pathogen burden in stool samples. Cognitive assessments will be completed at 2, 5, and 7 years of follow-up. The investigators hypothesize that children in households given the ceramic disk or the water filter will show improved linear growth compared to those in households without these interventions. The investigators expect that the ceramic disk will perform similarly to the water filter and result in similar improvements in linear growth when compared to children from control households.

Estimates of effectiveness demonstrated in this trial will provide the necessary evidence base to support the scale-up of manufacturing and distribution of the ceramic disks and filters, which could provide a robust point-of-use water treatment solution for rural areas. By helping to identify effective tools to reduce the risk of stunting in children, the trial will contribute to targets to improve child health in low-resource settings.

ELIGIBILITY:
Inclusion Criteria:

* Mother is in third trimester of pregnancy or there is at least one child under 3 years of age in the household
* The child's caregiver is at least 16 years of age

Exclusion Criteria:

* The household has chlorinated water piped into the home or routinely delivered (via truck or diversion) to a permanent, engineered system that stores the water within the property
* The household currently uses a ceramic filter or other commercial water treatment technology (including a permanent, engineered system that treats the water through filtration and/or chlorination)
* The household has plans to move outside the community in the next 6 months
* The youngest child under 3 years of age is seriously ill (has a severe disease requiring prolonged hospitalization or a severe or chronic condition diagnosed by medical doctor, e.g. neonatal disease, renal disease, chronic heart failure, liver disease, cystic fibrosis, congenital conditions)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 415 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Change in height-for-age z-score (ΔHAZ) | From 0-2 years of follow-up
  Height measured quarterly among all children under age 15 in the households, z-scores calculated from World Health Organization growth standards

SECONDARY OUTCOMES:
Change in weight-for-age z-score (ΔWAZ) | From 0-2 years of follow-up
  Weight measured quarterly among all children under age 15 in the households, z-scores calculated from WHO growth standards
Pathogen burden in stool samples | Quarterly from 0-2 years of follow-up
  Non-diarrheal stools collected from the youngest child under 3 years of age in each household; testing for enteroaggregative Escherichia coli, enterohemorrhagic Escherichia coli/EPEC, enterotoxigenic Escherichia coli, Shigella/enteroinvasive Escherichia coli, Giardia, Campylobacter, Cryptosporidium, Adenovirus by quantitative polymerase chain reaction
Prevalence of diarrhea | Quarterly from 0-2 years of follow-up
  7-day recall of diarrhea in the youngest child under 3 years of age in each household
Cognitive function - Bayley Scales of Infant Development III (ages 2-3); Wechsler Preschool and Primary Scale of Intelligence III (ages 3-6); Raven's Combined Matrices (ages > 6) | 2, 5, and 7 years of follow-up
  Cognitive assessments will be completed for the youngest child in each household (determined at enrollment) using age-appropriate developmental tests that have already been adapted, translated, and piloted in this population. Caregivers will be asked to bring their child to the local health clinic to be assessed by a Psychological Research Assistant.
Silver levels in treated water samples | Quarterly from 0-2 years of follow-up
  Treated water samples will be taken from a random subset of 50 households receiving the filter or ceramic disk every three months to determine the silver levels in treated water from the households. Total silver concentration will be measured by graphite furnace atomic absorption spectrometry (U.S.E.P.A. Method 7010).

CONTACTS AND LOCATIONS:
Overall Officials: Pascal O Bessong, PhD, Principal Investigator — University of Venda, Limpopo, South Africa; Rebecca Dillingham, MD, MPH, Principal Investigator — University of Virginia
Locations (1):
- University of Venda, Thohoyandou, Limpopo, South Africa

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Commercial website describing the main experimental device in this trial — http://madidrop.com/